CLINICAL TRIAL: NCT01741064
Title: Secondary Hyperparathyroidism Related Vascular and Bone Morbidity After Renal Transplantation - a 6 Year Follow up Retrospective Cohort Study.
Brief Title: Morbidity Related to Secondary Hyperparathyroidism After Renal Transplantation
Acronym: SHPT-RT
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Gunnar Sterner, MD, Ass. Prof, Skane University Hospital
Other Study IDs: SHPTTX-002
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Secondary Hyperparathyroidism; Disorder Related to Renal Transplantation
Keywords: Secondary Hyperparathyroidism; Renal Transplantation; Myocardial Infarction; Fracture; Graft Failure
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Myocardial Infarction; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PTH below target iPTH in CKD: iPTH at one year post transplantation below target range of iPTH by stage of CKD (KDOQI-guidelines).
- iPTH within target range of iPTH in CKD: iPTH at one year post transplantation within target range of iPTH by stage of CKD (KDOQI-guidelines).
- iPTH above target range of iPTH in CKD: iPTH at one year post transplantation above target range of iPTH by stage of CKD (KDOQI-guidelines).

SUMMARY:
The purpose of the study is to evaluate the long term vascular morbidity and mortality in kidney transplant recipients based on one year post transplant levels of intact parathyroid hormone.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism (SHPT) is a well known complication to chronic renal failure. With impaired renal function the phosphate excretion from the kidney is reduced. Together with low levels of 25- and 1,25-vitamin D3 and hypocalcemia this uremic mineral milieu drives the release of parathyroid hormone (PTH) and the development of SHPT. PTH has many functions but acts mainly to release calcium from the skeleton, to enhance calcium uptake from the intestines (by actions on vitamin D) and to lower serum phosphate by inducing phosphaturia. SHPT has been shown to cause vascular morbidity and fractures in the chronic kidney disease (CKD) patient. After successful renal transplantation (RT) the mineral disturbances are mostly recovered and stabilized at one year post RT, but in recent years it has been shown that SHPT persists in the major part of RT-recipients even after long term follow up. This has been associated with high risk of fractures and vascular related morbidity in the post transplant period. It has also been shown that low levels of iPTH in the post-transplant period might be associated with a high risk of fractures. Because of insufficient data on PTH levels and associated morbidity there is no specific recommendations of target PTH levels in the RT-patient. This indicates that there is need for further observational studies to describe the SHPT-associated morbidity in a post transplant cohort based on stabilized levels of post transplant iPTH.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-85 years at date of transplantation
* Signed informed consent or deceased at time of data collection

Exclusion Criteria:

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent renal transplantation surgery between January 1:st 2003 to December 31:st 2005 at Skane University Hospital or Karolinska University Hospital.
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
First Vascular Event | From date of transplantation to event up to 72 months
  Vascular events defined as (Myocardial infarction, Stroke, Peripheral Vascular Occlusion)

SECONDARY OUTCOMES:
Loss of Graft Function | From date of transplantation to event up to 72 months
  Start in Active Uremic Treatment (dialysis, renal transplantation)
Overall Mortality | Fram date of transplantation to event up to 72 months
  Mortality

OTHER OUTCOMES:
First Fracture | From date of transplantation to event up to 72 months
  Fracture verified by x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Sterner, MD A/Prof, Study Director — Dept of Nephrology and Transplantation Skane University Hospital Malmo; Astrid Seeberger, PhD, A/Prof, Study Chair — ´Dept of nephrology, Karolinska University Hospital Huddinge, Stockholm; Elin Isaksson, MD, Study Chair — Dept of Nephrology and Transplantation Skane University Hosptial Malmö

REFERENCES:
- [Background] Isaksson E, Sterner G. Early development of secondary hyperparathyroidism following renal transplantation. Nephron Clin Pract. 2012;121(1-2):c68-72. doi: 10.1159/000342811. Epub 2012 Oct 27. PMID 23107897
- [Background] Kanaan N, Claes K, Devogelaer JP, Vanderschueren D, Depresseux G, Goffin E, Evenepoel P. Fibroblast growth factor-23 and parathyroid hormone are associated with post-transplant bone mineral density loss. Clin J Am Soc Nephrol. 2010 Oct;5(10):1887-92. doi: 10.2215/CJN.00950110. Epub 2010 Jul 15. PMID 20634326
- [Background] Goldsmith D, Kothawala P, Chalian A, Bernal M, Robbins S, Covic A. Systematic review of the evidence underlying the association between mineral metabolism disturbances and risk of fracture and need for parathyroidectomy in CKD. Am J Kidney Dis. 2009 Jun;53(6):1002-13. doi: 10.1053/j.ajkd.2009.02.010. PMID 19463763
- [Background] Evenepoel P, Meijers BK, de Jonge H, Naesens M, Bammens B, Claes K, Kuypers D, Vanrenterghem Y. Recovery of hyperphosphatoninism and renal phosphorus wasting one year after successful renal transplantation. Clin J Am Soc Nephrol. 2008 Nov;3(6):1829-36. doi: 10.2215/CJN.01310308. Epub 2008 Oct 15. PMID 18922992